CLINICAL TRIAL: NCT03868280
Title: Fracture Table vs. Lateral Positioning for Intramedullary Fixation of Femur Fractures (The FLiP Study): A Pilot Cluster Randomized Crossover Trial
Brief Title: The FLiP Study, a Pilot Cluster Randomized Trial
Acronym: FLiP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Hamilton Academic Health Sciences Organization (Other); Canadian Orthopaedic Trauma Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CTO 2108
Record Dates: First submitted 2019-02-05; First posted 2019-03-11 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Femur Fracture
MeSH Terms: conditions — Femoral Fractures

STUDY DESIGN:
Intervention Model Description: Pilot cluster randomized crossover trial design
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supine Positioning, Fracture Table (Active Comparator): During the supine fracture table phase, patients will be positioned supine on a fracture table. The operative leg will be placed in a boot, attached to the traction limb. The non-operative leg will either be scissored away from the operating area in a traction boot (without traction placed) or placed in a stirrup at 90 degrees of hip flexion in hemi-lithotomy. A central post will be used to prevent patient movement during application of traction, and all bony prominences will be padded. Fluoroscopy will be obtained through standard practices intraoperative to document assessment of rotation.
  Interventions: Procedure: Antegrade femoral nailing Supine Position
- Lateral Positioning, Free drape (Active Comparator): During the lateral positioning phase, patients will be placed in lateral position after anaesthetic has been provided. A beanbag will be placed below the patient, and the patient will be safely turned to a lateral position. The beanbag will be inflated, the leg will be prepped, and a free drape will be applied. No traction will be used. Alternatively, some participating sites may use stulberg positioners rather than an inflatable beanbag, based on hospital preference. This positioning mirrors the positioning utilized for the direct lateral, posterior or posterolateral approach to a total hip arthroplasty or hemiarthroplasty
  Interventions: Procedure: Antegrade Femoral Nailing Lateral Position

INTERVENTIONS:
Procedure: Antegrade femoral nailing Supine Position — Antegrade femoral nailing in Supine Position using a Fracture Table
  Arms: Supine Positioning, Fracture Table
Procedure: Antegrade Femoral Nailing Lateral Position — Antegrade femoral nailing in Lateral Position using a Free drape
  Arms: Lateral Positioning, Free drape

SUMMARY:
The primary objective of this pilot trial is to assess the feasibility of a definitive trial to determine the effect of lateral patient positioning versus supine positioning with fracture table use for reamed antegrade intramedullary fixation of femur fractures.

DETAILED DESCRIPTION:
Femoral shaft fractures typically occur alongside other complex, high-energy injuries in the poly-traumatized patient. Femur fractures can cause extensive bleeding and surrounding muscle injury, and have a high global burden; occurring at a rate between 14 and 42.5 /100,000 person years, with approximately 1 in 10 road traffic accidents worldwide resulting in a femoral shaft fracture requiring surgery. Additionally, there is significant disparity in the burden of diaphyseal femur fractures, with 91% occurring in lower middle-class income countries, and the majority affecting younger males.

To help mitigate the effects of ongoing pain, blood-loss, worsening inflammation from unstable fracture ends, femoral shaft fractures require urgent management using either an early total-care or damage-control orthopaedics approach. Associated injuries, markers of resuscitation, and overall patient stability guide operative decision making and the timing of surgical intervention. Definitive internal fixation using reamed, locked intramedullary nailing (IMN) has become the standard of care in an adequately resuscitated patient, as it provides fracture stability while facilitating nursing care and patient mobilization. Multiple femoral IMN techniques exist; however, most femoral shaft fractures can be treated with an antegrade nail using either supine (fracture table) or lateral (free-leg drape) positioning.

Femoral Malrotation is a Common and Significant Complication

Despite the adoption of femoral IMN, patient-reported function following femur fracture fixation varies widely. Incorrect positioning of the fracture fragments by more than 15° relative to the native limb rotation (femoral malrotation) is associated with poor functional recovery, low health-related quality of life, gait abnormalities, difficulty with stairs, and delayed return to pre-injury activity. Significant femoral malrotation (>15°) occurs in up to 55% of patients following femoral shaft fracture IMN, as measured by post-operative computer tomography (CT) scans. Numerous intraoperative assessments have been used to judge rotation, including cortical diameter, lesser trochanter profile and others; though none are easily reproducible or reliable. The preferred technique by surgeons is the lesser trochanter profile, but this method requires a true anteroposterior view of the pelvis, which can be challenging to obtain with the fracture table in place.

A Lack of Consensus On Operative Table and Patient Positioning While the orthopaedic surgery community agrees that femoral shaft fractures should be treated with IMN, there is a lack of agreement on whether the patient should be placed in the supine position on fracture table (SFT) or in the lateral position on a standard radiolucent operating table (LRT). Our research team recently conducted a survey of the Canadian Orthopaedic Association membership and found a clear divide on patient positioning, with 56% of respondents using supine position on fracture table and 44% using a form of lateral positioning.

A recent comprehensive review identified only three studies on this specific topic. The best existing evidence of the previous literature comes from a prospective randomized trial led by Stephen et al. The authors described that supine positioning without use of fracture table yielded better post-operative rotation than patients treated with a fracture table. However, this study did not assess the utility of lateral positioning, which is more commonly used in isolated femoral shaft fractures. Moreover, the study was unable to associate malrotation with patient important outcomes or gait abnormalities. This clearly leaves much uncertainty surrounding optimal patient positioning during the definitive treatment of these critical injuries.

Proponents of positioning femoral shaft fracture patients using SFT argue that the fracture table provides a constant traction force to stabilize the fractured limb and allows for better intraoperative imaging. This arguably allows surgeons to reduce operative time and minimize the need for surgical assistants. However, possible downsides of this technique include the need for more invasive surgical adjuncts if there is ongoing difficulty with fracture reduction. Furthermore, constant and prolonged traction poses known risks to neurovascular structures associated with the central post, and may overpower feedback from the natural resting tone of the surrounding thigh musculature, possibly leading to a higher incidence of fixation in a malrotated position. Additionally, fracture tables are expensive and require additional setup in the operating room prior to the procedure.

Orthopedic surgeons who prefer the LRT believe it offers improved access to the start point for IMN as well as to the rest of the femur for manipulation, resulting in a better reduction of the fractured limb. With the entire limb free of traction, the thigh sits in a relatively adducted position at rest and the soft tissues tend to fall away from the operative field. The fracture fragments can be readily accessed and freely manipulated, with muscles returning to their resting tension as alignment is restored. It is believed that this leads to leads to improved limb alignment and less malrotation. Furthermore, there may be benefits to the overall patient, many of whom have other severe injuries that may also be impacted by intraoperative positioning. A recent cohort study, which was adjusted for associated injuries, found that patients treated using the LRT had shorter ICU stays and reduced number of days on a ventilator, indicating that there may be a protective effect from a respiratory standpoint. Additionally, the standard operating room table is readily available, less expense, and does not require additional setup prior to the procedure. However, there are concerns that lateral positioning may lead to longer operative times as additional positioning aids and reduction maneuvers may be required. Specifically, patients receiving delayed fixation may pose a challenge due to increased muscle shortening and tone that may be difficult to overcome with manual traction alone.

Limited previous studies align with biomechanical principles, and suggest that lateral positioning holds potential to reduce the incidence of femoral malrotation and avoid complications associated with the use of a fracture table; leading to improved patient function. Addressing malrotation by using the LRT may represent a simple and reproducible intervention that may improve quality of life for the patient.

NEED FOR A TRIAL Currently, the choice between the two techniques is dependent on surgeon preference, with very limited evidence to guide decision making. A large definitive trial is needed to answer this question and allow orthopaedic surgeons to make an evidence-based decision on how to treat patients with femoral shaft fractures, while reducing the incidence of malrotation and improving patient outcomes. Prior to embarking on a large definitive cluster randomized crossover trial (CRXO), a pilot study is needed to demonstrate feasibility. A pilot study would assess areas of uncertainty that may impact feasibility to perform the definitive trial, including achieving adequate recruitment, adherence to protocol, and minimal contamination.

ELIGIBILITY:
Inclusion Criteria:

1. Adult aged 18 years or older
2. Mid shaft (Diaphyseal) femur fracture appropriate for antegrade fixation
3. Surgery performed by participating surgeon or delegate
4. Provision of informed consent
5. Enrolled within 3 weeks of femoral shaft fixation

Exclusion Criteria:

• 1. Ipsilateral tibial fracture 2. Bilateral femur fracture 3. Ipsilateral femoral neck fracture 4. Ipsilateral acetabular fracture 5. Periprosthetic fracture 6. Pathologic fracture 7. Previous external fixation of femoral shaft fracture 8. Inability to be positioned in lateral decubitus because of a concomitant injury 9. Pregnancy (due to decubitus positioning) 10. Incarceration 11. Expected injury survival of less than 6 months 12. Terminal illness with expected survival of less than 6 months (expected follow up of study) 13. Inability to provide informed consent (e.g. cognitive disability, language barrier, significant delirium or dementia) 14. Currently involved in study that does not permit co-enrolment 15. Likely problems, in the judgment of study personnel, with maintaining follow-up with the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-10-16 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility to conduct definitive Clinical Trial | Six Months
  Our primary outcome for the pilot trial is feasibility, which includes the following:
  * Recruitment (number of participants recruited across all sites over study period, goal of approximately 100 participants)
  * Cluster crossover randomization protocol adherence
  * Complete primary outcome collection (CT scans) on all enrolled patients.
  * Participant retention and follow-up data
  * Accuracy of 15 degrees as a cut off for malrotation

SECONDARY OUTCOMES:
Postoperative femur alignment | Within 6 weeks of injury
  Immediate (within 6 weeks of surgery) post-operative bilateral computer tomography (CT scan) of the operated patients' lower extremity will be obtained as per standard of care. Postoperative bilateral CT scans for femoral shaft fractures represents the standard of care across academic centres(13). A physician familiar with musculoskeletal imaging, who is blinded to treatment allocation, will evaluate every CT for each participant. The best available literature defines clinically significant malrotation as more than 15 degrees difference from the contralateral limb in either internal or external rotation (
Health Related Quality of Life | up to 6 months
  Health-related quality of life will be assessed with the EQ-5D. The EQ-5D (27) questionnaire will be completed by participants at the time of consent and will ask about their pre-injury health status, as well as health status at the six weeks, three and six months follow up visits. The EQ-5D score represents patient reported health-related quality of life in five domains. The EQ-5D may be administered in person, over the telephone, standard mail, or electronically.
Modified Harris Hip Score | up to 6 months
  The modified Harris Hip Score is a limb specific functional score, which has been validated for use in other orthopedic populations, including those with total joint arthroplasty and hip fractures. The questionnaire will be completed by participants at each follow up appoints. The mHHS may be administered in person, electronically or by telephone.
Operative Time, Fluoroscopy Time | At time of Surgery
  Operative time will be defined as the time from induction of anaesthetic and ending once the patient has procedural wounds closed, documented through operative room records. Fluoroscopy time is defined as the total time that fluoroscopy is used and is recorded on the C-Arm used for intraoperative imaging. • The pain is in the study extremity
  * The pain began after surgery
  * The pain has persisted for at least three months after surgery
  * The pain is not better explained by an infection, malignancy, a pre-existing pain condition or any other alternative cause (as judged by the treating surgeon)
  * The severity of pain must be at least 4 on an 11-point NRS for average pain in the past week
Need for Open Reduction | At time of Surgery
  Need for open reduction is defined as any secondary incision at the fracture site >5 cm. This incision facilitates open reduction and is viewed as a surrogate measure of difficulty achieving the appropriate reduction using closed manipulation.
Use of Reduction Adjuncts | At time of Surgery
  Use of additional reduction adjuncts is defined as use of less invasive reduction aids (e.g. reduction clamps, joystick pins, F tool, and femoral distractor) not requiring a secondary incision (>5cm) at the fracture site
Operative Table Complications | At time of Surgery, Up to 6 months
  Standard operative table and fracture table complications include all potential neurological injuries (e.g. pudendal, peroneal and femoral nerve palsies, etc.) and skin injuries (e.g. skin blisters, ulceration, and skin tears, etc.) derived from use of the traction boot apparatus. These will also be documented in the medical record as per standard of care. Complications will be adjudicated by a blinded member of the study team, familiar with both the injury and nature of the operation.
Length of Hospital, ICU Stay | At initial admission
  Length of hospital stay will be defined as days from admission until the day of discharge to either home, rehabilitation care, or long-term care support. Days in ICU will be recorded according to medical records.
Days of Ventilator Support | At initial admission
  Days of ventilator support will be defined as discrete days spent receiving any form of positive pressure ventilation, including BiPAP while extubated.

CONTACTS AND LOCATIONS:
Overall Officials: Herman Johal, MD, Principal Investigator — McMaster University; Sheila Sprague, PhD, Principal Investigator — McMaster University; Daniel Axelrod, MD, Principal Investigator — McMaster University
Locations (3):
- Canada (2):
  - McMaster University, Hamilton, Ontario
  - Ottawa Civic Hospital, Ottawa, Ontario
- Vall d'Hebron University Hospital, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data will be available upon reasonable request to the Principal Investigators at the end of the study.
Supporting Information: Study Protocol
Time Frame: Data will be available for request at the end of the study, after primary publication has been completed.
Access Criteria: Requests will be reviewed by the Principal Investigators.